CLINICAL TRIAL: NCT01182974
Title: Paracetamol-induced Liver Toxicity in Septic Patients
Brief Title: Paracetamol Toxicity in Septic Patients
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty in patient enrollment
Sponsor: Barzilai Medical Center (Other)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Albert Grinshpun, Barzilai medical center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1662CTIL
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-03

CONDITIONS: Fever; Sepsis
Keywords: fever in severe sepsis
MeSH Terms: conditions — Fever; Sepsis | interventions — Acetaminophen; Dipyrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- paracetamol treatment (Active Comparator)
  Interventions: Drug: paracetamol
- control- dypirone treatment (Active Comparator)
  Interventions: Drug: dypirone

INTERVENTIONS:
Drug: paracetamol — 1 gr of paracetamol PO/PZ/PR
  Other Names: acetaminophen, acamol
  Arms: paracetamol treatment
Drug: dypirone — 1 gr PO/PZ/PR/IM
  Other Names: optalgin
  Arms: control- dypirone treatment

SUMMARY:
The investigators will examine the toxicity of therapeutic doses of paracetamol in patients in severe sepsis. Patients with fever and severe sepsis will be randomized to receive paracetamol or dypirone. The investigators will monitor blood glutathione and liver enzymes to look for potential toxicity.

DETAILED DESCRIPTION:
Paracetamol is metabolized in liver using the glutathione system. This detoxification system is depressed during severe illness such as sepsis, trauma etc. The study will examine the toxicity of therapeutic doses of paracetamol in patients in severe sepsis. We believe that during sepsis, paracetamol metabolites are not fully detoxified and therefore are toxic to the patient.

Patients with fever and severe sepsis will be randomized to receive paracetamol or dypirone. The investigators will monitor blood glutathione (as a surrogate marker for liver glutathione), liver enzymes and various clinical data (such as length of hospitalization) to look for a potential toxicity.

ELIGIBILITY:
Inclusion Criteria:

* age>18y
* hospitalized to int. med. dept. or ICU
* body temp>38 and one or more from the following:

  1. pulse>90 bpm
  2. resp. rate>20/min or PaCO2<32 mmHg
  3. WBC>12000 or <4000
* one of the following:

  1. hypotension
  2. disturbed end-organ perfusion (confusion, oliguria, lactic acidosis etc.)

Exclusion Criteria:

* acute / chronic liver disease
* acute CNS disorder
* current isoniazid treatment
* alcoholism
* active malignancy
* pregnancy
* TPN or PPN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
paracetamol induced liver toxicity | every six months
  defined as ALT and/or AST > 1000 or reduction in glutathione below 50% of base line

CONTACTS AND LOCATIONS:
Overall Officials: Albert Grinshpun, Principal Investigator — Barziali medical center, Ashkelon
Locations (1):
- Barzilai medical center, Ashkelon, Israel